CLINICAL TRIAL: NCT05813600
Title: To Evaluate the Efficacy and Safety of Nirmatrelvir/Ritonavir in the Treatment of the Omicron Variant of COVID-19
Brief Title: Efficacy and Safety of Nirmatrelvir/Ritonavir for Treating Omicron Variant of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangao Jiang (Other)
Responsible Party: Sponsor-Investigator, Xiangao Jiang, Director, Wenzhou Central Hospital
Organization: Wenzhou Central Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Xiangao Jiang
Record Dates: First submitted 2023-04-07; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Omicron Variant of COVID-19
Keywords: Nirmatrelvir/Ritonavir; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lianhua qingwen granule (No Intervention): Patients were given Lianhua Qingwen Capsule orally, 3 times/day, 6 g/time. oral antipyretic (ibuprofen suspension 10ml) and symptomatic supportive treatment for body temperature >38.5 ℃.
- lianhua qingwen granule+Nirmatrelvir/Ritonavir (Experimental): Patients were given Lianhua Qingwen Capsule orally, 3 times/day, 6 g/time. oral antipyretic (ibuprofen suspension 10ml) and symptomatic supportive treatment for body temperature >38.5 ℃. And given Nirmatrelvir 300mg/Ritonavir 100mg orally, q12h, for 5 days.
  Interventions: Drug: Nirmatrelvir/Ritonavir

INTERVENTIONS:
Drug: Nirmatrelvir/Ritonavir — Patients in both groups were given Lianhua Qingwen Capsule orally, 3 times/day, 6 g/time. oral antipyretic (ibuprofen suspension 10ml) and symptomatic supportive treatment for body temperature >38.5 ℃. The study group was given Nirmatrelvir 300mg/Ritonavir 100mg orally, q12h, for 5 days, and the control group not given any antiviral drugs.
  Arms: lianhua qingwen granule+Nirmatrelvir/Ritonavir

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Nirmatrelvir/Ritonavir in the treatment of the Omicron variant of COVID-19. The main question it aims to answer is: Whether the use of the drug can help patients recover from COVID-19.

Patients in both groups were given Lianhua Qingwen Capsule orally, 3 times/day, 6 g/time. oral antipyretic (ibuprofen suspension 10ml) and symptomatic supportive treatment for body temperature >38.5 ℃. The study group was given Nirmatrelvir 300mg/Ritonavir 100mg orally, q12h, for 5 days, and the control group not given any antiviral drugs.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of COVID-19 infection within 24h and positive nasopharyngeal swab for COVID-19 nucleic acid RNA；
* Age ≥12 years and weight ≥ 40Kg；
* Subjects of fertility must agree to use highly effective contraceptive methods.

Exclusion Criteria:

* Previous history of COVID-19 treatment；
* The known history of active liver disease；
* Patients on renal dialysis or have moderate to severe impaired renal function；
* The known human immunodeficiency virus (HIV) infection;
* Suspected or confirmed concurrent active systemic infections other than COVID-19 infection；
* Allergy or other contraindication to any component of the study intervention;
* Any drug or substance that is currently or expected to be used that is a high reliance on CYP3A4 enzyme clearance or strong CYP3A4 enzyme inducers；
* pregnant or breastfeeding women.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-08 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Nasal swab COVID-19 nucleic acid tests | On days 4, 7, 9 and 11 of treatment
  Patients in both groups underwent nasal swab COVID-19 nucleic acid tests on days 4, 7, 9 and 11 of treatment, and CT values were recorded (CT values of 40 for negative results). Compare the difference in the change of CT values of COVID-19 nucleic acid between two groups of patients
Virus turn negative | From date of randomization until the date of first documented progression, assessed up to 5 months
  Compare the first negative conversion(or CT value ≥35) time of coronavirus nucleic acid between two groups
Hospital stays | From date of randomization until the date of first documented progression, assessed up to 5 months
  Compare the difference in hospitalization time between the two groups strictly according to discharge criteria
Adverse drug reaction | From date of randomization until the date of first documented progression, assessed up to 5 months
  Compare the adverse drug reactions during hospitalization between two groups
COVID-19 nucleic acid re-positive | From date of randomization until the date of first documented progression, assessed up to 5 months
  After discharge, patients in both groups continued to be isolated at the isolation point for 7 days and underwent COVID-19 nucleic acid tests daily to compare the COVID-19 nucleic acid re-positive

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangao Jiang, Wenzhou, Zhejiang, China